CLINICAL TRIAL: NCT03539406
Title: Intraperitoneal Infusion of ex Vivo-cultured Allogeneic NK Cells in Recurrent Ovarian Carcinoma Patients (a Phase I Study)
Brief Title: Intraperitoneal Infusion of ex Vivo-cultured Allogeneic NK Cells in Recurrent Ovarian Carcinoma Patients
Acronym: INTRO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL60937.000.17
Record Dates: First submitted 2018-02-12; First posted 2018-05-29 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2022-10

CONDITIONS: Recurrent Ovarian Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: This study is a phase I safety and feasibility study in a series of 12 patients who are suffering from recurrent ovarian, fallopian tube or primary peritoneal cancer. The first cohort of three patients will receive an intraperitoneal infusion of allogeneic UCB-NK cells generated ex vivo from CD34+ hematopoietic progenitor cells obtained from an allogeneic UCB unit without a preparative regimen. In the second group of three patients the same UCB-NK cell dosage will be given with a preparative regimen of four days non-myeloablative immunosuppressive conditioning regimen with cyclophosphamide and fludarabine (CyFlu). If no severe toxicity is seen in these 6 patients, an extension cohort of 6 patients will be included to answer the secondary objective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NK-cells without preparative regimen (Experimental): NK-cells without preparative regimen
  Interventions: Biological: UCB-NK cells
- NK-cells with preparative regimen (Experimental): NK-cells with preparative regimen
  Interventions: Biological: UCB-NK cells; Drug: Chemotherapy

INTERVENTIONS:
Biological: UCB-NK cells — Intraperitoneal allogeneic UCB-NK cells infusion
Drug: Chemotherapy — Cyclofosfamide/fludarabine treatment
  Arms: NK-cells with preparative regimen

SUMMARY:
This study investigates an innovative treatment for recurrent ovarian cancer exploiting ex vivo-generated allogeneic natural killer (NK) cells with or without preceding non-myeloablative conditioning chemotherapy.

DETAILED DESCRIPTION:
This study investigates an innovative treatment for recurrent ovarian cancer exploiting ex vivo-generated allogeneic natural killer (NK) cells with or without preceding non-myeloablative conditioning chemotherapy.

This study is a phase I safety and feasibility study in a series of 12 patients who are suffering from recurrent ovarian, fallopian tube or primary peritoneal cancer. Prior to NK cell infusion, a laparoscopy is performed to place a catheter in the peritoneal cavity. The first cohort of three patients will receive an intraperitoneal infusion of allogeneic UCB-NK cells generated ex vivo from CD34+ hematopoietic progenitor cells obtained from an allogeneic UCB unit without a preparative regimen. In the second group of three patients the same UCB-NK cell dosage will be given with a preparative regimen of four days non-myeloablative immunosuppressive conditioning regimen with cyclophosphamide and fludarabine (CyFlu). If no severe toxicity is seen in these 6 patients, an extension cohort of 6 patients will be included to answer the secondary objective.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from their second recurrence of ovarian, fallopian tube or primary peritoneal cancer, with an elevated serum level of CA-125 on two successive time points with 28 days in between, reaching a value of more than 2 times nadir and above 35 U/ml without gastrointestinal symptoms.
* Able to undergo laparoscopic IP port placement and IP treatment administration
* Adequate organ function
* Age 18 years or older
* Age under 76 years.
* Karnofsky performance status >70% (see appendix 2)
* Life expectancy > 6 months
* At least 28 days after last anti cancer treatment, before start of preparative regimen
* Written informed consent
* Availability of a partially HLA-matched UCB unit

Exclusion Criteria:

* Patients on immunosuppressive drugs
* Patients with active infections (viral, bacterial or fungal) that requires specific therapy. Acute anti-infectious therapy must have been completed within 14 days prior to study treatment
* Laparoscopic adhesion score >4 out of 9.
* Severe cardiovascular disease (arrhythmias requiring chronic treatment, congestive heart failure or symptomatic ischemic heart disease (appendix 4)
* Severe pulmonary dysfunction (CTCAE III-IV) (appendix 4)
* Severe renal dysfunction (MDRD<50) (appendix 4)
* Severe hepatic dysfunction (serum bilirubin or transaminases > 3 times normal level) (appendix 4)
* Severe neurological or psychiatric disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 6 months
  Incidence of treatment emergent adverse events (following CTCAE criteria)

SECONDARY OUTCOMES:
in vivo lifespan of the infused UCB-NK cells | 28 days
  determination of NK cell percentage in blood and peritoneal fluid
in vivo expansion of the infused UCB-NK cells | 28 days
  determination of NK cell percentage in peritoneal fluid and blood
Measurement of in vitro cytolytic activity of infused NK cells | 28 days
  in CFSE base killing assays a percentage of dead cells (K562 cells) will be measured.
the effect of NK cell infusion on measurable disease | 6 months
  CA-125 testing in blood (in E/mL)
the effect of NK cell infusion on measurable disease | 6 months
  CT-scan (measurement of visible leasions in cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No